CLINICAL TRIAL: NCT00176631
Title: A Phase II Trial of Licorice Root and Docetaxel in Patients With Hormone Refractory Prostate Cancer
Brief Title: Licorice Root Extract and Docetaxel in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000539682; P30CA072720 (NIH); 0220034593 (Other: UMDNJ IRB); CINJ 080306 (Other: CINJ)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Glycyrrhiza glabra extract; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- licorice root extract and docetaxel (Experimental)
  Interventions: Dietary Supplement: licorice root extract; Drug: docetaxel

INTERVENTIONS:
Dietary Supplement: licorice root extract — Licorice root is started on Day 1 and is given at a dose of 6.75 g each day (five 450 mg capsules tid) for a total of 21 days in each cycle.
Drug: docetaxel — All the patients will be treated with docetaxel at a dose of 60 mg/m2 every 21 days on Day 1 of the treatment cycle.

SUMMARY:
RATIONALE: Licorice root extract contains ingredients that may slow the growth of tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving licorice root extract together with docetaxel may be an effective treatment for prostate cancer.

PURPOSE: This phase II trial is studying the side effects and how well giving licorice root extract together with docetaxel works in treating patients with metastatic prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and toxicity of licorice root extract in combination with docetaxel in patients with hormone-refractory metastatic prostate cancer.

Secondary

* Determine the ability of licorice root extract to alter surrogate markers of estrogen activity and cytotoxicity in these patients.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1 and oral licorice root extract 3 times a day on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate adenocarcinoma

  * Metastatic disease
* Must have failed initial hormonal therapy and have disease progression after at least one chemotherapy regimen*, meeting any of the following criteria:

  * Progressive PSA ≥ 5 ng/mL, as evidenced by 2 separate measurements taken ≥ 2 weeks apart with the second PSA measurement greater than the first one and PSA measurement at screening greater than the first one
  * Progressive measurable disease (e.g., changes in the size of lymph nodes or parenchymal masses or appearance of new lesions on physical examination or x-ray/CT scan) with a PSA level at screening ≥ 5 ng/mL
  * Progressive bone metastasis (e.g., presence of new lesions on a bone scan) with a PSA level at screening ≥ 5 ng/mL NOTE: *Prior chemotherapy must include a taxane therapy, but disease progression does not have to follow taxane therapy
* Patients must maintain primary androgen ablation (hormonal) therapy AND experience disease progression while not receiving antiandrogen therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,500/mm^3
* Bilirubin ≤ 1.2 mg/dL
* Creatinine ≤ 1.5 mg/dL
* SGOT or SGPT ≤ 1.5 times upper limit of normal
* No other prior malignancy unless treated with curative intent and free of disease for the time period considered appropriate for the specific cancer
* No uncontrolled hypertension
* No active infections
* No known HIV positivity
* No uncontrolled medical condition that would preclude study therapy
* No diagnosis of major depression or suicidal ideation
* No problems with oral absorption

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior surgery or radiotherapy and recovered
* At least 4 weeks since prior flutamide
* At least 6 weeks since prior bicalutamide
* No prior or concurrent herbal supplements or thiazide diuretics
* No other concurrent investigational or commercial agents or therapies

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. DiPaola, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://www.clinicaltrials.gov/ct2/show/NCT00176631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten subjects were enrolled from April 2004 through November 2006 at Rutgers Cancer Institute of New Jersey, a comprehensive cancer center, and one of its affiliate hospitals within the CINJ Oncology Group.
Groups:
- Licorice Root Extract and Docetaxel: licorice root extract : Licorice root is started on Day 1 and is given at a dose of 6.75 g each day (five 450 mg capsules tid) for a total of 21 days in each cycle.
  docetaxel : All the patients will be treated with docetaxel at a dose of 60 mg/m2 every 21 days on Day 1 of the treatment cycle.
Period: Overall Study
Arm/Group | Licorice Root Extract and Docetaxel
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Licorice Root Extract and Docetaxel
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With PSA Response
Description: Decline from baseline value by > 50%, or normalization of PSA (defined as PSA less than 0.2 ng/ml), confirmed by a second measurement at least 1 or more weeks later.
Time Frame: 9 months
Population: No data collected
Arm/Group | Licorice Root Extract and Docetaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Patients With a Decrease in BCL-2 Levels in PBMC and in the Degree of Plasma ER Receptor, Between Patients Who Responded to Treatment and Patients Who Did Not
Time Frame: 9 months
Population: No data collected
Arm/Group | Licorice Root Extract and Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Licorice Root Extract and Docetaxel
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Licorice Root Extract and Docetaxel (N=10)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Licorice Root Extract and Docetaxel (N=10)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 8 (11)
Constitutional Symptoms - Other (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (22)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (24)
Hemoglobin (Blood and lymphatic system disorders) | 3 (6)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (2)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (2)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Bone pain (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (Cardiac disorders) | 3 (3)
Hypotension (Cardiac disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Auditory/Hearing - Other (Ear and labyrinth disorders) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (2)
Hypermagnesemia (Investigations) | 1 (1)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes